CLINICAL TRIAL: NCT04818489
Title: Impact of Colchicine on the Clinical Outcome of COVID-19 and the Development of Post-COVID-19 Pulmonary Fibrosis: Randomized Controlled Clinical Trial
Brief Title: Colchicine and Post-COVID-19 Pulmonary Fibrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ClinAmygate (Other)
Responsible Party: Principal Investigator, Emad R Issak, Doctor, ClinAmygate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR00202
Record Dates: First submitted 2021-02-13; First posted 2021-03-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Pulmonary Fibrosis Interstitial
Keywords: COVID19; Pulmonary Fibrosis; Colchicine; Clinical outcomes
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis | interventions — Colchicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiologist who will assess the CT scans will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine group (Experimental): Colchicine 0.5 mg (2 tablets: 1 mg) twice per day as a loading dose, followed by one tablet 0.5 twice per day for three weeks in addition to the local standard protocol of COVID19 management
  Interventions: Drug: Colchicine 0.5 MG; Other: the standard protocol only
- Control group (Placebo Comparator): the local standard protocol of COVID19 management
  Interventions: Other: the standard protocol only

INTERVENTIONS:
Drug: Colchicine 0.5 MG — colchicine 0.5 mg (2 tablets: 1 mg) twice per day as a loading dose, followed by one tablet 0.5 twice per day for three weeks in addition to the standard protocol
  Other Names: Colchicine
  Arms: Colchicine group
Other: the standard protocol only — the local standard protocol for COVID19
  Other Names: the local standard protocol for COVID19

SUMMARY:
Pulmonary fibrosis is a sequela to adult respiratory distress syndrome (ARDS). 40% of patients with corona virus disease 2019 (COVID-19) develop ARDS, and 20% of them are severe. Clinical, radiographic, and autopsy reports of pulmonary fibrosis were commonplace following SARS and MERS, and current evidence suggests pulmonary fibrosis could complicate infection by SARS-CoV-2 too. Colchicine has a direct anti-inflammatory effect by inhibiting the synthesis of tumor necrosis factor alpha and IL-6, monocyte migration, and the secretion of matrix metalloproteinase-9. It suppress secretion of cytokines and chemokines as well as in vitro platelet aggregation. All these are potentially beneficial effects that might diminish the COVID-19 inflammatory storm associated with severe cases.

DETAILED DESCRIPTION:
Approximately 96 million people have been diagnosed with severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), and around two million people have died from this deadly disease worldwide. The pulmonary symptoms associated with SARS-CoV-2 vary from mild respiratory symptoms to severe respiratory failure. Of those infected with SARS-CoV-2, 40% will progress to ARDS.

Radiologically, most of those infected by SARS COV 2 have bilateral lower lobes ground-glass opacities with or without consolidation. However, long term lung impairment may develop particularly interstitial lung disease (ILD), the fibrotic type. Besides, pulmonary fibrosis (PF) is recognized sequelae of ARDS, and several studies have shown that protective lung ventilation tends to diminish the radiographic abnormalities following ARDS.

Colchicine has anti-fibrotic effects as a microtubule-destabilizing agent. In an in vitro study using human lung fibroblasts, colchicine inhibited myofibroblast differentiation via Rho/serum response factor (SRF) dependent. In COVID19 cases, colchicine was used by where they assessed its impact on the inflammatory biomarkers and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are confirmed to have COVID-19 clinically, radiologically and PCR
* Age above 18 years old
* Informed written consent

Exclusion Criteria:

* History of hypersensitivity to colchicine
* Pregnancy or breastfeeding women.
* Patients with severe renal impairment (creatinine clearance (CCL) <30 mL / min)
* Patients with severe hepatic impairment (AST or ALT> 5 times the normal limits in International Units (ULN)
* Patients with blood dyscrasias, neutrophils <1.000 / mmc or platelets <50.000 / mmc
* Patients with history of severe cardiac insufficiency
* Patients with history of pulmonary fibrosis
* Severe diarrhoea or bowel diverticulitis, or perforation
* Patients who cannot take oral therapy
* Patients already in ICU or requiring mechanical ventilation
* Patients already enrolled in other clinical trials
* Patients with taking P-glycoprotein inhibitor (e.g. ciclosporin, verapamil or quinidine) or a CYP3A4 inhibitor (e.g. ritonavir, remdesivir, atazanavir, indinavir, clarithromycin, telithromycin, itraconazole or ketaconazole) or Tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Clinical status | Two weeks
  Seven-category ordinal scale: minimum 1 is the best and a maximum is 6
Pulmonary fibrosis at week 2 | Two weeks
  Percent of Participants with pulmonary fibrosis
Pulmonary fibrosis at 45 days | 45 days
  Percent of Participants with pulmonary fibrosis

SECONDARY OUTCOMES:
C-reactive protein | Two weeks
  Change in the levels of C-reactive protein
Ferritin | Two weeks
  Change in the levels of Ferritin
Erythrocyte sedimentation rate | Two weeks
  Change in the levels of Erythrocyte sedimentation rate
Lactate dehydrogenase | Two weeks
  Change in the levels of Lactate dehydrogenase
Adverse events | 45 days
  Adverse events related to the study medication
Pulmonary function test: FVC | 45 days
  Pulmonary function test: FVC
Pulmonary function test: FEV1 | 45 days
  Pulmonary function test: FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Emad Issak, Principal Investigator — Ain Shams Univeristy
Locations (1):
- El-Demerdash Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deftereos SG, Giannopoulos G, Vrachatis DA, Siasos GD, Giotaki SG, Gargalianos P, Metallidis S, Sianos G, Baltagiannis S, Panagopoulos P, Dolianitis K, Randou E, Syrigos K, Kotanidou A, Koulouris NG, Milionis H, Sipsas N, Gogos C, Tsoukalas G, Olympios CD, Tsagalou E, Migdalis I, Gerakari S, Angelidis C, Alexopoulos D, Davlouros P, Hahalis G, Kanonidis I, Katritsis D, Kolettis T, Manolis AS, Michalis L, Naka KK, Pyrgakis VN, Toutouzas KP, Triposkiadis F, Tsioufis K, Vavouranakis E, Martinez-Dolz L, Reimers B, Stefanini GG, Cleman M, Goudevenos J, Tsiodras S, Tousoulis D, Iliodromitis E, Mehran R, Dangas G, Stefanadis C; GRECCO-19 investigators. Effect of Colchicine vs Standard Care on Cardiac and Inflammatory Biomarkers and Clinical Outcomes in Patients Hospitalized With Coronavirus Disease 2019: The GRECCO-19 Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e2013136. doi: 10.1001/jamanetworkopen.2020.13136. PMID 32579195
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014